CLINICAL TRIAL: NCT01505881
Title: Evaluation of the Long Term Safety of the Use of Dabigatran Etexilate in Patients With a Bileaflet Mechanical Heart Valve
Brief Title: Follow on Study From RE-ALIGN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1160.138; 2011-002285-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Thromboembolism; Heart Valve Prosthesis
MeSH Terms: conditions — Thromboembolism | interventions — Dabigatran; Warfarin

ARMS (2):
- Dabigatran etexilate (Experimental): Patient dose determined by dose allocated in 1160.113 and CrCl levels
  Interventions: Drug: dabigatran etexilate low dose; Drug: dabigatran etexilate intermediate dose; Drug: dabigatran etexilate high dose
- warfarin (Active Comparator): warfarin doses to maintain INR levels
  Interventions: Drug: warfarin 5mg; Drug: warfarin 1mg; Drug: warfarin 3mg

INTERVENTIONS:
Drug: dabigatran etexilate low dose — active treatment (low)
  Arms: Dabigatran etexilate
Drug: warfarin 5mg — comparator warfarin
  Arms: warfarin
Drug: dabigatran etexilate intermediate dose — active treatment (medium)
  Arms: Dabigatran etexilate
Drug: warfarin 1mg — comparator warfarin
  Arms: warfarin
Drug: dabigatran etexilate high dose — active treatment (high)
  Arms: Dabigatran etexilate
Drug: warfarin 3mg — comparator warfarin
  Arms: warfarin

SUMMARY:
To collect additional data relating to safety and indicators of efficacy for patients who have participated in the 1160.113 study.

ELIGIBILITY:
Inclusion criteria:

1. Completed study 1160.113 per protocol
2. Continuing need for anticoagulation

Exclusion criteria:

1. uncontrolled hypertension
2. severe renal impairment
3. active liver disease
4. increased risk of bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (30):
- Belgium (3):
  - 1160.138.32003 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.138.32002 Boehringer Ingelheim Investigational Site, Genk
  - 1160.138.32001 Boehringer Ingelheim Investigational Site, Leuven
- Canada (5):
  - 1160.138.11001 Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - 1160.138.11009 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.138.11011 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1160.138.11012 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1160.138.11007 Boehringer Ingelheim Investigational Site, Toronto, Ontario
- Czechia (4):
  - 1160.138.42002 Boehringer Ingelheim Investigational Site, Brno
  - 1160.138.42003 Boehringer Ingelheim Investigational Site, Olomouc
  - 1160.138.42004 Boehringer Ingelheim Investigational Site, Ostrava
  - 1160.138.42001 Boehringer Ingelheim Investigational Site, Prague
- Denmark (2):
  - 1160.138.45001 Boehringer Ingelheim Investigational Site, Copenhagen
  - 1160.138.45002 Boehringer Ingelheim Investigational Site, Odense C
- France (4):
  - 1160.138.33004 Boehringer Ingelheim Investigational Site, Bron
  - 1160.138.33001 Boehringer Ingelheim Investigational Site, Paris
  - 1160.138.33002 Boehringer Ingelheim Investigational Site, Pessac
  - 1160.138.33003 Boehringer Ingelheim Investigational Site, Rennes
- Germany (5):
  - 1160.138.49001 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.138.49002 Boehringer Ingelheim Investigational Site, Essen
  - 1160.138.49004 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1160.138.49003 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1160.138.49010 Boehringer Ingelheim Investigational Site, Witten
- Netherlands (2):
  - 1160.138.31002 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.138.31004 Boehringer Ingelheim Investigational Site, Breda
- Norway (2):
  - 1160.138.47002 Boehringer Ingelheim Investigational Site, Bergen
  - 1160.138.47001 Boehringer Ingelheim Investigational Site, Oslo
- Poland (3):
  - 1160.138.48004 Boehringer Ingelheim Investigational Site, Gdansk
  - 1160.138.48003 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.138.48001 Boehringer Ingelheim Investigational Site, Wroclaw

REFERENCES:
- [Derived] Eikelboom JW, Connolly SJ, Brueckmann M, Granger CB, Kappetein AP, Mack MJ, Blatchford J, Devenny K, Friedman J, Guiver K, Harper R, Khder Y, Lobmeyer MT, Maas H, Voigt JU, Simoons ML, Van de Werf F; RE-ALIGN Investigators. Dabigatran versus warfarin in patients with mechanical heart valves. N Engl J Med. 2013 Sep 26;369(13):1206-14. doi: 10.1056/NEJMoa1300615. Epub 2013 Aug 31. PMID 23991661

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran Etexilate (DE): Oral administration of 1 capsule of 150 mg (150 mg), 2 capsules of 110 mg (220 mg), or 2 capsules of 150 mg (300 mg) twice daily.
- Warfarin: Oral administration of Warfarin 1mg, 3mg and 5 mg according to target international normalised ratio (INR), as recommended in guidelines, and deemed appropriate by investigator
Period: Overall Study
Arm/Group | Dabigatran Etexilate (DE) | Warfarin
Started | 99 | 59
Completed | 95 | 58
Not Completed | 4 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TRT): The TRT comprised all patients who were documented to have taken at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate (DE) | Warfarin | Total
Number analyzed (Participants) | 99 | 59 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (8.0) | 56.1 (10.1) | 57.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 19 | 56
  Male | 62 | 40 | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Any Adverse Event (AE)
Description: Percentage of patients with Adverse Events. Prespecified clinical outcome events were not recorded as Adverse Events.
Time Frame: From first intake of study drug until last intake of study drug plus 6 days (Up to 272 days)
Population: Treated set (TRT): The TRT comprised all patients who were documented to have taken at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate (DE) | Warfarin
Number analyzed (Participants) | 99 | 59
percentage of participants | 39.4 | 37.3

2. Secondary Outcome: Percentage of Patients With AEs Leading to Discontinuation of Trial Drug
Description: Percentage of patients with Adverse Events leading to discontinuation of trial drug.
  Prespecified clinical outcome events were not recorded as Adverse Events.
Time Frame: From first intake of study drug until last intake of study drug plus 6 days (Up to 272 days)
Population: Treated set (TRT): The TRT comprised all patients who were documented to have taken at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate (DE) | Warfarin
Number analyzed (Participants) | 99 | 59
percentage of participants | 5.1 | 1.7

3. Secondary Outcome: Percentage of Patients With Serious AEs
Description: Percentage of patients with Serious Adverse Events (SAE). Prespecified clinical outcome events were not recorded as Adverse Events.
Time Frame: From first intake of study drug until last intake of study drug plus 6 days (Up to 272 days)
Population: Treated set (TRT): The TRT comprised all patients who were documented to have taken at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate (DE) | Warfarin
Number analyzed (Participants) | 99 | 59
percentage of participants | 3.0 | 6.8

4. Secondary Outcome: Percentage of Deaths, Venous Thromboembolism (VTE), Myocardial Infarction (MI), Transient Ischaemic Attacks (TIA), Strokes, Systemic Embolism, and Valve Thrombosis.
Description: Clinical efficacy outcome events presented are:
  Death, Venous thromboembolism (VTE), Myocardial Infarction (MI), Transient Ischaemic Attack (TIA), Stroke, Systemic embolism and Valve thrombosis
Time Frame: From first intake of study drug until last intake of study drug plus 6 days (Up to 272 days)
Population: Treated set (TRT): The TRT comprised all patients who were documented to have taken at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate (DE) | Warfarin
Number analyzed (Participants) | 99 | 59
percentage of participants
  Death | 0.0 | 1.7
  Venous thromboembolism | 0.0 | 0.0
  Myocardial Infarction | 1.0 | 0.0
  Transient Ischaemic Attack | 1.0 | 0.0
  Stroke | 3.0 | 0.0
  Systemic embolism | 0.0 | 0.0
  Valve thrombosis | 2.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first intake of study drug until last intake of study drug plus 6 days (Up to 272 days)
Description: Patients are presented according to the treatment they received except for 2 patients, who mistakenly switched to study warfarin during the study. These patients are presented under the Dabigatran columns only.
Groups:
- Dabigatran Etexilate: Oral administration of 1 capsule of 150 mg (150 mg), 2 capsules of 110 mg (220 mg), or 2 capsules of 150 mg (300 mg) twice daily
Arm/Group | Dabigatran Etexilate | Warfarin
Serious Adverse Events (participants affected / at risk) | 3/99 | 4/59
Other Adverse Events (participants affected / at risk) | 5/99 | 4/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (N=99) | Warfarin (N=59)
Cellulitis (Infections and infestations) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (N=99) | Warfarin (N=59)
Hypertension (Vascular disorders) | 5 | 4

LIMITATIONS AND CAVEATS:
This study was terminated prematurely due to safety concerns arising during conduct of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.